CLINICAL TRIAL: NCT04948034
Title: A Phase Ⅱ Trial of Multisite Stereotactic Ablative Radiotherapy (SABR) Combined With Fruquintinib and Tislelizumab in Metastatic Colorectal Cancer
Brief Title: The Combination of Fruquintinib, Tislelizumab and Stereotactic Ablative Radiotherapy in Metastatic Colorectal Cancer(RIFLE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2020-274-2194
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A total of 68 metastatic colorectal cancer patients who have failed the first-line standard treatment will receive multisite SABR followed by Fruquintinib and Tislelizumab within two weeks from completion.
  The dosing of Tislelizumab will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR); Drug: Fruquintinib; Drug: Tislelizumab

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — We plan to irradiate as many metastatic lesions as possible, in the precondition that normal tissues can tolerate.
  Target dose will be adjusted depending on site of the lesion and organs at risk (BED > 100Gy).
  Treatment schedule is once per day and five days per week. Sequence of irradiation for multiple metastases is at the discretion of the investigators based on their experience.
Drug: Fruquintinib — Starts within two weeks upon SABR completion: 5mg, d1-14, qd; Continued until disease progression, unacceptable toxicity or patient withdrawal.
Drug: Tislelizumab — Starts within one week upon SABR completion: 200mg, d1, q3w; the dosing will continue for up to two years until disease progression, unacceptable toxicity or patient withdrawal.

SUMMARY:
This is a prospective, single-center, single-arm phase II clinical trial.This study aims to evaluate the safety and tolerability of stereotactic ablative radiotherapy (SABR) in combination with Fruquintinib and Tislelizumab, and to examine the impact of the combination therapy on tumor control, long-term survival and quality of life in patients with Metastatic colorectal cancer.

A total of 68 metastatic colorectal cancer patients who have failed the first-line standard treatment, will be recruited and receive multisite SABR(8-12 Gy, 4-5 times) followed by fruquintinib(5mg, qd) and tislelizumab(200mg, q3w) within two weeks from completion.The overall response rate (ORR), disease control rate(DCR), progression-free survival(PFS) and overall survival(OS) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old, regardless of gender
* Fully informed and willing to provide written informed consent for the trial
* ECOG performance status 0-1
* Has an investigator determined life expectancy of at least 6 months
* Histologically or cytologically confirmed stage IV colorectal cancer (UICC 8th version)
* Has at least 2 measurable oligometastatic lesions on imaging (RECIST version 1.1). One will be treated with SABR and the other will be biopsied and evaluated against RECIST 1.1.
* Has progressive disease after receiving first-line standard antitumor therapy (chemotherapeutic agents including fluorouracil, oxaliplatin and irinotecan); previous neoadjuvant or adjuvant pelvic area radiotherapy is allowed; subjects included in the safety introduction phase may include third-line treatment or above, but these subjects will not be included in the final statistical analysis.
* Subjects receiving adjuvant oxaliplatin should progress during adjuvant therapy or within 6 months after completion.
* Demonstrate adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.
* Subjects who withdraw from standard treatment before disease progressing due to unacceptable toxicity and exclude the use of the same drug are also allowed to be included.
* Non pregnant or lactating patients. Effective contraceptive methods should be used during the study and within 6 months of the last administration.

Exclusion Criteria:

* Pregnant or lactating women
* The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years excluding adequately treated non-melanoma skin cancer, carcinoma in situ of cervix and superficial bladder tumor (non-invasive tumor, or carcinoma in situ, or T1)
* Baseline laboratory indicators do not meet the following criteria: neutrophils ≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L , ALT ≤2.5 ULN, AST ≤2.5 ULN, Cr≤ 1.5 ULN or creatinine clearance rate <50ml/min, TBIL ≤1.5 ULN, APTT ≤1.5 ULN, PT ≤1.5 ULN (the criteria of patients with liver metastasis: PLT ≥80×10^9/L, ALT ≤5 ULN, AST ≤5 ULN, TBIL ≤2.5 ULN)
* Serious electrolyte abnormalities
* Urinary protein ≥ 2+, or 24-hour urine protein ≥1.0g/24h
* Uncontrolled hypertension: SBP >140mmHg or DBP > 90mmHg
* Receiving radiotherapy within 4 weeks
* Receiving anti-VEGF or anti-EGFR therapy within 4 weeks
* Stroke event or transient ischemic attack occurred within 12 months
* A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months
* A histroy of heart disease within 6 months (including congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting, cardiac insufficiency ≥ NYHA grade 2 and LVEF<50%)
* Uncontrolled malignant pleural effusion, ascites, or pericardial effusion
* Previous treatment with immunotherapy or fruquintinib
* The presence of gastrointestinal diseases such as gastric or duodenal active ulcers, ulcerative colitis or unresected tumors with active bleeding; or other conditions likely to cause gastrointestinal bleeding or perforation; or unhealed gastrointestinal perforation or gastrointestinal fistula after surgical treatment
* A history of liver disease including, but not limited to HBV infection or HBV DNA positive(≥1×10^4/ml), HCV infection or HCV DNA positive(≥1×10^3/ml) and liver cirrhosis
* Serious mental abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years
  The percentage of patients with objective response in the non-irradiated metastatic lesions. Objective response is defined as complete response (CR) or partial response (PR) per response evaluation criteria (RECIST v1.1) and the immune related response criteria (iRECIST) after treatment.

SECONDARY OUTCOMES:
Disease Control Rate | Up to 2 years
  The percentage of patients with disease control in the non-irradiated metastatic lesions. Disease control is defined as CR, PR, or stable disease (SD) per RECIST v1.1 and iRECIST after treatment.
Duration of Response | Up to 2 years
  Defined as the time between PR/CR and subsequent progression disease (PD) per RECIST v1.1 and iRECIST or death from any cause.
Progression-Free Survival | Up to 3 years
  Defined as the time from initiation of treatment to PD or death from any cause.
Overall Survival | Up to 3 years
  Defined as the time from initiation of treatment to death from any cause.
Acute Toxicity | Up to 2 years
  The percentage of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang K, Chen Y, Zhang Z, Wu R, Zhou M, Yang W, Wan J, Shen L, Zhang H, Wang Y, Han X, Wang J, Zhang Z, Xia F. RIFLE: a Phase II trial of stereotactic ablative radiotherapy combined with fruquintinib and tislelizumab in metastatic colorectal cancer. Gastroenterol Rep (Oxf). 2023 Oct 11;11:goad063. doi: 10.1093/gastro/goad063. eCollection 2023. PMID 37842200